CLINICAL TRIAL: NCT01280929
Title: Prospective, Randomized, Multicenter, Open Label, Phase II Study to Access Efficacy and Safety of Lucentis® Monotherapy (Ranibizumab 0.5 mg Intravitreal Injections) Compared With Lucentis® Plus Panretinal Photocoagulation (PRP) and PRP (Monotherapy) in the Treatment of Patients With High Risk Proliferative Diabetic Retinopathy
Brief Title: Prospective, Randomized, Multicenter, Open Label, Phase II Study to Access Efficacy and Safety of Lucentis® Monotherapy Compared With Lucentis® Plus Panretinal Photocoagulation (PRP) and PRP in the Treatment of Patients With High Risk Proliferative Diabetic Retinopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: José Cunha-Vaz (Other)
Responsible Party: Sponsor-Investigator, José Cunha-Vaz, Investigator Coordinator, Association for Innovation and Biomedical Research on Light and Image
Organization: Association for Innovation and Biomedical Research on Light and Image (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002DPT04T; 2009-014409-15 (EudraCT Number)
Record Dates: First submitted 2011-01-20; First posted 2011-01-21 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: High Risk Proliferative Diabetic Retinopathy
Keywords: High Risk Proliferative Diabetic Retinopathy; Ranibizumab; Panretinal Photocoagulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Panretinal Photocoagulation (PRP) (Active Comparator): Group 1: Panretinal photocoagulation treatment (PRP) at month-0 that can be repeated after month-3.
  Interventions: Procedure: Panretinal Photocoagulation (PRP)
- Ranibizumab (Experimental): Group 2: Intravitreous injections of ranibizumab every 4 weeks at month-0, month-1 and month-2 that can be repeated after month-3.
  Interventions: Drug: Intravitreous injection of ranibizumab
- Ranibizumab + Panretinal Photocoagulation (PRP) (Experimental): Group 3: Combination treatment of ranibizumab intravitreous injections plus PRP (2 weeks +/- 1 week after injection), at month-0, month-1 and month-2 that can be repeated after month-3.
  Interventions: Procedure: Panretinal Photocoagulation (PRP); Drug: Intravitreous injection of ranibizumab

INTERVENTIONS:
Procedure: Panretinal Photocoagulation (PRP)
  Arms: Panretinal Photocoagulation (PRP); Ranibizumab + Panretinal Photocoagulation (PRP)
Drug: Intravitreous injection of ranibizumab
  Arms: Ranibizumab; Ranibizumab + Panretinal Photocoagulation (PRP)

SUMMARY:
The purpose of this trial is to evaluate safety and to compare the efficacy of intravitreous injection of ranibizumab alone (0.5 mg), versus combination of intravitreous injection of ranibizumab (0.5 mg) plus panretinal photocoagulation, versus panretinal photocoagulation alone in the regression of retinal neovascularization in eyes with high-risk proliferative diabetic retinopathy.

DETAILED DESCRIPTION:
Panretinal photocoagulation can cause regression of retinal neovascularization and reduce the risk of severe vision loss in people with proliferative diabetic retinopathy. However, this destructive treatment may be associated with side effects (such as: pain, transient blurring, loss of peripheral and/or night vision, increased risk of macular edema and central vision loss) and it is not always efficient in the regression of the neovascularization.

Vascular endothelial growth factor (VEGF) has been shown to play a role in retinal neovascularization and retinal vascular leakage related with proliferative diabetic retinopathy and diabetic macular edema. Anti-vascular endothelial growth factor treatments have been hypothesized as an alternative adjunctive treatment for the management of retinal neovascularization and macular edema related with diabetic retinopathy.

There are a few reports of retinal traction detachment in patients with proliferative diabetic retinopathy and fibrovascular proliferation (although it is not frequent). However, from our clinical experience, we think that the risk of detachment only exists when there is in place a fibrovascular proliferation with retinal traction previous to the injection.

We injected ranibizumab prior to surgery in patients with severe proliferative diabetic retinopathy, that were submitted later to a posterior vitrectomy, to reduce neovascularization and minimize the risk of an intraoperatory hemorrhage caused by the manipulation of the fibrovascular membranes. In total, we already injected and submitted to surgery 15 eyes with the above mentioned condition, with excellent results. The results of the first 10 eyes were presented in the congress of the Portuguese Society of Ophthalmology (2008).

ELIGIBILITY:
Inclusion Criteria:

* High-risk proliferative diabetic retinopathy (HR-PDR) eyes.
* Best Corrected-Visual Acuity at baseline > 20/320 in the study eye.
* Clear ocular media and adequate pupillary dilatation to permit good quality fundus photography.
* Intraocular pressure < 21 mmHg.
* Type I, or Type II diabetic subjects as defined by the World Health Organization criteria of either gender, and aged ≥ 18 years.
* Women must be using effective contraception, be post-menopausal for at least 12 months prior to trial entry, or surgically sterile.
* Ability to provide written informed consent.
* Ability to return for all trial visits.

Exclusion Criteria:

* Eyes with prior scatter (panretinal) or focal/grid photocoagulation, within the previous 6 months.
* Fibrovascular proliferation with retinal traction.
* Other cause of retinal neovascularization (retinal vein occlusion, radiation retinopathy or others).
* Atrophy/scarring/fibrosis/ hard exudates involving the center of the macula.
* Subjects who have received yttrium-aluminum-garnet laser, or peripheral retinal cryoablation, or laser retinopexy (for retinal tears only), or focal/grid photocoagulation, within the previous 6 months.
* Significant media opacities, which might interfere with visual acuity, assessment of toxicity or fundus photography.
* Subjects should not be entered if there is likelihood that they will require cataract surgery within the following 1 year.
* Any intraocular surgery within 6 months before trial enrollment.
* Previous vitrectomy.
* HbA1C level >11% or recent signs of uncontrolled diabetes.
* Any of the following underlying systemic diseases:

  * History or evidence of severe cardiac disease.
  * History or evidence of clinically significant peripheral vascular disease such as intermittent claudication or prior amputation.
  * Clinically significant impaired renal function (serum creatinine >2.5 mg/dL or s/p renal transplant or receiving dialysis).
  * Clinically significant impaired hepatic function.
  * Stroke (within 12 months of trial entry).
  * Any major surgical procedure within one month before trial enrollment.
* Previous radiation to the head in the region of the study eye.
* Any prior treatment with an investigational agent for diabetic retinopathy or anti-VEGF therapy (including intravitreal, subconjunctival or subtenons corticosteroids) during the past 90 days for any other condition.
* Known serious allergies to fluorescein used in angiography, or to components of Lucentis® formulation.
* Systolic Blood Pressure > 170 (2 different readings) or diastolic Blood Pressure > 100 (2 different readings).
* Acute ocular or periocular infection.
* Previous filtering surgery (e.g., trabeculectomy) or placement of a glaucoma drainage device (e.g., tube-shunt surgery).
* Use of other investigational drugs at the time of enrollment.
* History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes.
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL).
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant UNLESS they are: women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner; women whose partners have been sterilized by vasectomy or other means using a highly effective method of birth control. Periodic abstinence are not acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Regression of neovascularization | 12-month treatment
  To demonstrate superiority of one of the treatment arms: ranibizumab 0.5 mg monotherapy, panretinal photocoagulation monotherapy or combination therapy (ranibizumab 0.5 mg plus panretinal photocoagulation) over a 12-month treatment period in the regression of neovascularization.

SECONDARY OUTCOMES:
Changes from baseline in Best-Corrected Visual Acuity | 12-month treatment
  Best-Corrected Visual Acuity will be assessed during the trial (Baseline, Month 3, Month 6 and Month 12).
Changes from baseline in macular retinal thickness by Optical Coherent Tomography | 12-month treatment
  Optical Coherent Tomography will be assessed during the trial (Baseline, Month 3, Month 6 and Month 12).
Recurrence of neovascularization | 12-month treatment
  To assess if there is recurrence of neovascularization.
Number of treatments needed | 12-month treatment
  To analyse the number treatments given to each subject during the the 12-month treatment.
Additional focal or grid laser for Diabetic Macular Edema | 12 month treatment
  To assess the number of patients that received additional focal or grid laser for Diabetic Macular Edema.
Adverse events | 12-month treatment
  Drug safety profile.
Need for vitrectomy due to occurrence of vitreous hemorrhage or retinal detachment relative to the three treatment arms. | 12-month treatment
  To assess the number of subjects who needed vitrectomy due to occurrence of vitreous hemorrhage or retinal detachment relative to the three treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: José Cunha-Vaz, MD, PhD, Study Chair — Association for Innovation and Biomedical Research on Light and Image; João Figueira, MD, Principal Investigator — Center for Clinical Trials - Association for Innovation and Biomedical Research on Light and Image
Locations (7):
- Portugal (7):
  - Center for Clinical Trials - Association for Innovation and Biomedical Research on Light and Image, Coimbra
  - Espaço Médico de Coimbra, Coimbra
  - ALM Oftalmolaser, Lisbon
  - Instituto de Retina de Lisboa, Lisbon
  - Instituto de Oftalmologia Dr. Gama Pinto, Lisbon
  - Instituto CUF, Porto
  - Hospital de São João, Porto

REFERENCES:
- [Derived] Figueira J, Silva R, Henriques J, Caldeira Rosa P, Lains I, Melo P, Goncalves Nunes S, Cunha-Vaz J. Ranibizumab for High-Risk Proliferative Diabetic Retinopathy: An Exploratory Randomized Controlled Trial. Ophthalmologica. 2016;235(1):34-41. doi: 10.1159/000442026. Epub 2015 Dec 3. PMID 26630400